CLINICAL TRIAL: NCT05031702
Title: Effectiveness of the Assumption of a Supplement Based on the Extract From Camelia Leaf Sinensis on Basal Metabolism and Body Composition in Overweight Women or With Obesity in Postmenopause
Brief Title: Camelia Sinensis for Basal Metabolism and Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0905/14122018
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-08

CONDITIONS: Postmenopausal Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator): Extract from Camellia Sinensis leaf
  Interventions: Dietary Supplement: Camellia Sinensis leaf extract
- Placebo (Placebo Comparator): Tablets of the same size as the active component
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: Camellia Sinensis leaf extract — 2 tablets per day of 150 mg (1 before lunch and 1 before dinner)
  Arms: Dietary supplement
Combination Product: Placebo — 2 tablets per day of 150 mg (1 before lunch and 1 before dinner)
  Arms: Placebo

SUMMARY:
Camellia Sinensis leaf extract contributes to increasing energy expenditure and calorie consumption by increasing thermogenesis. The purpose of this study is to evaluate the efficacy of Camellia Sinensis on basal metabolism and body composition in overweight women or with obesity in postmenopause.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopause
* Overweight or obesity class I-II (Body Mass Index 25-39,9 Kg/m2)

Exclusion Criteria:

* Changes in heart rhythm
* Intolerance or allergy to components
* Obesity class III (Body Mass Index > 40 Kg/m2)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Changes on energy expenditure | Changes from baseline energy expenditure at 4 and at 8 weeks
  Basal metabolic rate (Kcal/day)
Changes on energy expenditure | Changes from baseline energy expenditure at 4 and at 8 weeks
  24 h urinary nitrogen (g/24 h)

SECONDARY OUTCOMES:
Changes on body composition | Changes from baseline body composition at 4 and at 8 weeks
  Fat Free Mass (g), Fat Mass (g), Visceral Adipose Tissue (g)
Changes on anthropometry | Changes from baseline anthropometry at 4 and at 8 weeks
  Weight (kg)
Changes on anthropometry | Changes from baseline anthropometry at 4 and at 8 weeks
  Body Mass Index (kg/m2)
Changes on anthropometry | Changes from baseline anthropometry at 4 and at 8 weeks
  Waist circumference (cm)
Changes on insulin resistance | Changes from baseline insulin resistance at 4 and at 8 weeks
  Homeostasis Model Assessment (pt) for evaluate insulin resistance if > 2,4
Changes on carbohydrate profile | Changes from baseline carbohydrate profile at 4 and at 8 weeks
  Glycemia (mg/dl)
Changes on carbohydrate profile | Changes from baseline carbohydrate profile at 4 and at 8 weeks
  Insulin (mcIU/ml)
Changes on lipid profile | Changes from baseline lipid profile at 8 weeks
  Total Cholesterol (mg/dl), High Density Lipoprotein Cholesterol (mg/dl), Low Density Lipoprotein Cholesterol (mg/dl), Tryglicerides (mg/dl)
Changes on inflammation | Changes from baseline inflammation at 8 weeks
  C-Reactive Protein (mg/dl)
Changes on incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline incidence of Treatment-Emergent Adverse Events at 8 weeks
  Alanine Aminotrasferase (IU/l), Aspartate Aminotrasferase (IU/I)
Changes on incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline incidence of Treatment-Emergent Adverse Events at 8 weeks
  Gamma Glutamyl Trasferase (U/l)
Changes on citokine profile | Changes from baseline citokine profile at 4 and at 8 weeks
  Adiponectin (microg/ml)
Changes on citokine profile | Changes from baseline citokine profile at 4 and at 8 weeks
  Leptin (ng/ml)
Changes on plasma catecholamine profile | Changes from baseline plasma catecholamine profile at 4 and at 8 weeks
  Adrenalin (ng/ml), Noradrenalin (ng/ml)
Changes on satiety | Changes of satiety through 8 weeks
  Haber test (pt) for evaluation of satiety from 0 (no satiety) to 10 (a lot of satiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Mariangela Rondanelli, Pavia, Italy